CLINICAL TRIAL: NCT04187612
Title: Association of Body Fluid Distribution with Obstructive Sleep Apnea in Pregnant Women with Body Mass Index ≥ 40 Kg/m2 - a Prospective Observational Study
Brief Title: Association of Body Fluid Distribution with Obstructive Sleep Apnea in Pregnant Women with Body Mass Index ≥ 40 Kg/m2
Status: Active, not recruiting | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 19-06
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Apnea, Obstructive Sleep; Obesity
Keywords: pregnancy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Total body water measurement: Total body water will be measured using Bioelectrical Impedance Analysis (BIA).
  Interventions: Device: Bioelectrical Impedance Analysis (BIA)

INTERVENTIONS:
Device: Bioelectrical Impedance Analysis (BIA) — BIA will be used to determine total body water

SUMMARY:
Obstructive Sleep apnea (OSA) is a common and underdiagnosed condition in obese pregnant women with serious and life-threatening complications to the mother and baby. The investiators propose that a non-invasive method may be used to detect patients at risk of OSA, giving these women access to the necessary treatment to treat this condition. The method is a estimation of body water, which has been shown to be linked to OSA in the non-pregnant population. Body water is estimated by applying surface electrodes to a participant who is lying down by measuring bioimpedance through body tissues by applying a tiny current between the electrodes. The electrical stimulation is not felt by the participant and has no negative effects on mother or baby.

DETAILED DESCRIPTION:
It is already established that the increasingly prevalent condition of obesity is linked to OSA in pregnancy. Obesity is increasingly prevalent This study will evaluate a novel method of screening for OSA in the obese pregnant population, thereby treating this condition reducing the ill effects to mother and fetus.

This will be a prospective observational cohort study. Eligible participants will be approached for consent during their third-trimester antenatal all-day clinic visit. Body water will be measured by connecting electrodes to participants hands, feet and neck whilst lying supine for approximately 15 minutes.

Data on patient demographics, BMI, medical conditions, water body composition and indicators of OSA (breathing pattern and oxygen levels during sleep) will be collected, as well as data from patients' sleep tests as ordered by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Participants who give written informed consent
* Pregnant women in the third trimester of pregnancy
* Grade III obesity
* Patients who have prior diagnosis of OSA within the last one year, and non-compliant to treatment such as continuous positive airway pressure (CPAP), or dental appliance
* Patients suspected to have OSA based on screening questionnaire (see page 2, OSA-Diagnostic tools for further details)

Exclusion Criteria:

* Fluid overload states including renal disease, liver disease and congestive heart failure
* Prior history of vascular surgery in the lower limbs such as varicose vein surgery, vascular by-pass surgery or evidence of venous efficiency.
* Patients with metal implants in lower limbs or spine, due to possible interference with the leg impedance signals. 58
* Participants with diagnosed OSA treated with Continuous Positive Airway Pressure (CPAP).
* Patients requiring urgent sleep physician referral (within four weeks) due to serious medical conditions or safety critical-occupations according to the 2011 Canadian Thoracic Society (CTS) guideline 59 e.g. unstable ischemic heart disease, recent cerebrovascular disease.
* Implantable cardiac devices

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Eligible participants will be approached for consent at our high risk maternal and infant program clinic on the day of their regularly scheduled appointment.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Presence of sleep apnea | 12 hours
  The diagnosis of sleep apnea will be made using apnea hypopnea index (AHI). A diagnosis of OSA is present if a person has an AHI ≥5/hour.

SECONDARY OUTCOMES:
Total body water measurement | Following consent, this measurement will be done, and will take approximately 30 minutes
  Total body water will be measured using Bioelectrical Impedance Analysis (BIA)
Mallampati score | Done during initial exam following consent, this exam will take 1-2 minutes
  The patient is asked to open their mouth wide and stick out their tongue. Upon observation, the view is classified/scored as Class 1-4. Class one would be least likely to have airway problems and 4 most likely.
Thyromental distance (cm) | Done during initial exam following consent, this exam will take 1-2 minutes
  The distance between the thyroid notch and the tip of the jaw with the head extended is evaluated.
Subluxation of mandible beyond maxilla | Done during initial exam following consent, this exam will take 1-2 minutes
  The patient is asked to extend their mandible beyond the top lip if possible. Scoring is yes or no.
Neck extension | Done during initial exam following consent, this exam will take 1-2 minutes
  The patient is asked to extend their neck, looking upwards and back, as far as comfortably possible. Scoring is yes if movement is possible, no if extension is not possible.
Height (cm) | Done during initial exam following consent, this exam will take 1-2 minutes
  Height measured in cm to calculate Body Mass index (BMI)
Weight (kg) | Done during initial exam following consent, this exam will take 1-2 minutes
  Weight measured in kg to calculate Body Mass index (BMI)
Neck size | Done during initial exam following consent, this exam will take 1-2 minutes
  Circumference around the neck, measured in centimeters.
Questionnaire related to snoring | Done during initial exam following consent, this exam will take 1-2 minutes
  Patients will be asked if they snore, if others can hear their snoring and if they are bothered by it. Yes or no answers.
Questionnaire related to sleep | Done during initial exam following consent, this exam will take 1-2 minutes
  Patients will be asked if they wake frequently during sleep, if they wake with a choking sensation, and whether they doze off or fall asleep while sitting/talking. Yes or no answers.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No